CLINICAL TRIAL: NCT04917757
Title: Clinical Outcome of Autonomous Cortisol Secretion in Adrenal Incidentalomas - Substudy of the ENSAT (European Network for the Study of Adrenal Tumor) Registry
Brief Title: Clinical Outcome of Autonomous Cortisol Secretion in Adrenal Incidentalomas
Acronym: NAPACA
Status: Active, not recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: European Network for the Study of Adrenal Tumors (Other Government)
Responsible Party: Principal Investigator, Martin Fassnacht, Chair Dept. of Endocrinology and Diabetes, Wuerzburg University Hospital
Other Study IDs: NAPACA-Outcome
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Adrenal Incidentaloma
MeSH Terms: conditions — Adrenal incidentaloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 1mg Dexamethasone test — For each patient a 1mg dexamethasone test has been performed.

SUMMARY:
The primary aim of the study is to assess mortality and cardiovascular events potentially linked to cortisol excess in patients with adrenal incidentalomas stratified by cortisol values following the 1-mg overnight dexamethasone test.

DETAILED DESCRIPTION:
The NAPACA Outcome Study is part of the ENSAT Registry (https://registry.ensat.org/)

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* adrenal incidentaloma (≥ 1cm) detected by cross-sectional imaging between January 1, 1996 and December 31, 2015
* imaging characteristics suggestive for an adrenal adenoma or excluded malignancy by follow-up imaging
* availability of a 1 mg dexamethasone test result
* follow-up data on living status and occurrence of cardiovascular events
* follow-up duration of at least 36 months.

Exclusion Criteria:

* proven pheochromocytoma, primary hyperaldosteronism or adrenocorticotropic hormone (ACTH)-dependent Cushing's syndrome
* clinical features suggestive for overt Cushing's syndrome; urinary free cortisol (UFC) ≥ 2-fold higher than the upper limit of normal of the local assay
* any active malignancy (including adrenocortical cancer) at the time of primary diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with adrenal incidentaloma
Sampling Method: Probability Sample
Enrollment: 3656 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fassnacht, MD, Study Chair — Wuerzburg University Hospital
Locations (2):
- University Hospital Würzburg, Würzburg, Germany
- University Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided.

REFERENCES:
- [Result] Deutschbein T, Reimondo G, Di Dalmazi G, Bancos I, Patrova J, Vassiliadi DA, Nekic AB, Debono M, Lardo P, Ceccato F, Petramala L, Prete A, Chiodini I, Ivovic M, Pazaitou-Panayiotou K, Alexandraki KI, Hanzu FA, Loli P, Yener S, Langton K, Spyroglou A, Kocjan T, Zacharieva S, Valdes N, Ambroziak U, Suzuki M, Detomas M, Puglisi S, Tucci L, Delivanis DA, Margaritopoulos D, Dusek T, Maggio R, Scaroni C, Concistre A, Ronchi CL, Altieri B, Mosconi C, Diamantopoulos A, Iniguez-Ariza NM, Vicennati V, Pia A, Kroiss M, Kaltsas G, Chrisoulidou A, Marina LV, Morelli V, Arlt W, Letizia C, Boscaro M, Stigliano A, Kastelan D, Tsagarakis S, Athimulam S, Pagotto U, Maeder U, Falhammar H, Newell-Price J, Terzolo M, Fassnacht M. Age-dependent and sex-dependent disparity in mortality in patients with adrenal incidentalomas and autonomous cortisol secretion: an international, retrospective, cohort study. Lancet Diabetes Endocrinol. 2022 Jul;10(7):499-508. doi: 10.1016/S2213-8587(22)00100-0. Epub 2022 May 6. PMID 35533704

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-functioning Adenoma: cortisol values after an overnight 1 mg dexamethasone suppression test; less than 50 nmol/L
- Adenoma With Possible Autonomous Cortisol Secretion: cortisol values after an overnight 1 mg dexamethasone suppression test: 50-138 nmol/L
- Adenoma With Autonomous Cortisol Secretion: cortisol values after an overnight 1 mg dexamethasone suppression test: > 138 nmol/L
Period: Overall Study
Arm/Group | Non-functioning Adenoma | Adenoma With Possible Autonomous Cortisol Secretion | Adenoma With Autonomous Cortisol Secretion
Started | 2089 | 1320 | 247
Completed | 2089 | 1320 | 247
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-functioning Adenoma | Adenoma With Possible Autonomous Cortisol Secretion | Adenoma With Autonomous Cortisol Secretion | Total
Number analyzed (Participants) | 2089 | 1320 | 247 | 3656
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1404 | 726 | 134 | 2264
  >=65 years | 685 | 594 | 113 | 1392
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [52 to 67] | 63 [52 to 67] | 63 [55 to 70] | 61 [53 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1321 | 860 | 169 | 2350
  Male | 768 | 460 | 78 | 1306
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 28 | 5 | 67
  Not Hispanic or Latino | 2011 | 1271 | 238 | 3520
  Unknown or Not Reported | 44 | 21 | 4 | 69
Region of Enrollment [Number; unit: participants]
  Europe | 154 | 98 | 18 | 270
  United States | 1935 | 1222 | 229 | 3386
adenoma diameter [Median (Inter-Quartile Range); unit: mm] | 20 [15 to 25] | 26 [19 to 33] | 29 [20 to 37] | 22 [15 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: death
Time Frame: From date of primary diagnosis of the adrenal incidentaloma to the date of death or last follow-up (data lock August 31, 2019). Median follow-up duration was 7.0 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-functioning Adenoma | Adenoma With Possible Autonomous Cortisol Secretion | Adenoma With Autonomous Cortisol Secretion
Number analyzed (Participants) | 2089 | 1320 | 247
Participants | 143 | 168 | 41

2. Secondary Outcome: Cardiovascular Morbidity
Description: Cardiovascular (CV) events (myocardial infarction, percutaneous coronary intervention, coronary bypass, stroke, deep vein thrombosis, and pulmonary embolism)
Time Frame: From date of primary diagnosis of the adrenal incidentaloma to the date of the first CV event or death or last follow-up (data lock August 31, 2019). Median follow-up duration was 7.0 years.
Population: The number of analyzed patients is slightly smaller than the total cohort, because for some patients no data on cardiovascular outcome were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-functioning Adenoma | Adenoma With Possible Autonomous Cortisol Secretion | Adenoma With Autonomous Cortisol Secretion
Number analyzed (Participants) | 1892 | 1208 | 225
Participants | 145 | 130 | 22

ADVERSE EVENTS:
Time Frame: From the date of primary diagnosis of the adrenal incidentaloma until the date of death or last follow-up (data lock December 31, 2018). Median follow-up duration was 7.0 years.
Description: Serious adverse events are defined major adverse cardiovascular events (MACE): myocardial infarction or coronary revascularisation (either bypass surgery or percutaneous intervention), stroke, or cardiovascular-related death.
  Time frame for MACE was defined as the time between the initial diagnosis of the adrenal incidentaloma and first documentation of any MACE thereafter.
Arm/Group | Non-functioning Adenoma | Adenoma With Possible Autonomous Cortisol Secretion | Adenoma With Autonomous Cortisol Secretion
All-Cause Mortality (participants affected / at risk) | 143/2089 | 168/1320 | 41/247
Serious Adverse Events (participants affected / at risk) | 145/1892 | 130/1208 | 22/225
Other Adverse Events (participants affected / at risk) | 724/2002 | 547/1250 | 123/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-functioning Adenoma (N=1892) | Adenoma With Possible Autonomous Cortisol Secretion (N=1208) | Adenoma With Autonomous Cortisol Secretion (N=225)
MACE (Cardiac disorders) | 145 | 130 | 22 — major adverse cardiovascular events (MACE): myocardial infarction or coronary revascularisation (either bypass surgery or percutaneous intervention), stroke, or cardiovascular-related death
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-functioning Adenoma (N=2002) | Adenoma With Possible Autonomous Cortisol Secretion (N=1250) | Adenoma With Autonomous Cortisol Secretion (N=232)
Dylipidemia (Metabolism and nutrition disorders) | 724 | 547 | 123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT04917757/Prot_SAP_000.pdf